CLINICAL TRIAL: NCT03357978
Title: Susceptibility to Infections, Tumor Risk and Liver Disease in Patients With Ataxia Telangiectasia With and Without Substitution of Immunoglobulin G: a Prospective Observational Study
Brief Title: Susceptibility to Infections, Tumor Risk and Liver Disease in Patients With Ataxia Telangiectasia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Stefan Zielen, Prof. Dr. med. Stefan Zielen, Johann Wolfgang Goethe University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: InfectionandLiver_AT2016
Record Dates: First submitted 2017-04-24; First posted 2017-11-30 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Ataxia Telangiectasia
Keywords: immunodeficiency; liver disease; cancer risk
MeSH Terms: conditions — Ataxia Telangiectasia; Immunologic Deficiency Syndromes; Liver Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A-T patients (Other): A-T patients aged 2 to 45 years with and without immunoglobulin G Substitution
  * bioelectrical impedance Analysis
  * blood draw
  * transient elastography (FibroScan)
  * ataxia score
  * Five-Times-Sit-to-Stand Test
  Interventions: Diagnostic Test: bioelectrical impedance analysis; Diagnostic Test: blood draw; Diagnostic Test: transient elastography (FibroScan); Diagnostic Test: ataxia score; Diagnostic Test: Five-Times-Sit-to-Stand Test

INTERVENTIONS:
Diagnostic Test: bioelectrical impedance analysis — Electrophysical measurement that allows to determine the exact composition of single body compartments by producing a magnetic field and detecting the potential difference through the body
Diagnostic Test: blood draw — Blood samples are taken from sober patients
Diagnostic Test: transient elastography (FibroScan) — FibroScan is a noninvasive tool to measure liver stiffness as an indication of fatty liver and liver fibrosis using ultrasound
Diagnostic Test: ataxia score — Klockgether ataxia score ranges from 0 to 35 points in which 0 means no symptoms and 35 stands for final stage of disease. It includes seven ataxia associated symptoms: dysarthria, intention tremor, ataxia of gait, stance, dysdiadochokinesia, upper limb and lower limb
Diagnostic Test: Five-Times-Sit-to-Stand Test — The test measures the complete time which is necessary for an individual to stand up and sit down on a chair five times in series

SUMMARY:
Ataxia telangiectasia (A-T) is a rare devastating human recessive disorder characterized by progressive cerebellar ataxia, immunodeficiency, chromosomal instability and cancer susceptibility. The immunodeficiency is expressed by recurring infections. It's characterised by decreased lymphocytes data as well as lack of immunglobulin A, immunglobulin G subclasses and specific antibodies against pneumococcus. Aim of the present clinical trial is to investigate frequency-, intensity- and duration of the infections as well as changes oft immune status, dimension of liver disease and tumor risk in patients with A-T, with and without immunoglobulin G substitution therapy. Transient elastography (FibroScan) will be performed in order to measure liver stiffness as an indication of fatty liver and liver fibrosis. A bioelectrical impedance analysis (BIA) is conducted to investigate the exact body composition. Ataxia Score is determined to define neurological problems. Every subject receives a diary to compile symptoms of infection.

DETAILED DESCRIPTION:
Ataxia teleangiectasia (A-T) is a rare devastating human recessive disorder characterized by progressive cerebellar ataxia, immunodeficiency, chromosomal instability and cancer susceptibility. The immunodeficiency is expressed by recurring infections. It's characterised by decreased lymphocytes data as well as lack of immunglobulin A, immunglobulin G subclasses and specific antibodies against pneumococcus as shown in many trials. Additionally the patients suffer from a fatty liver with increased transaminases and have the risk for a cirrhosis of the liver and a hepatocellular carcinoma. It's known that the dimension of the liver disease affects susceptibility to infection. Nevertheless there are only a few studies treating this problem.

Despite the proof of the immunodeficiency polyvalent immunoglobulins (IgG) are not given regularly. Own observations show that in spite of the treatment with immunoglobulins the progression of a chronic destructive lung disease with development of bronchiectasis hardly can prohibited.

Up to now it isn't cleared if a substitution therapy with immunoglobulins reduces the susceptibility to infection. Therefore the aim oft the present clinical trial ist to explore frequency-, intensity, and duration oft the infections as well as changes oft the immune status, measure of liver disease and tumor risk in patients with A-T, with and without immunoglobulin therapy. The study includes five visits, which are performed in all A-T patients. Visit 1, 3, 5 are realized in the context of annual follow ups:

* To evaluate weight and length of all subjects
* To analyze the exact structure of single body compartments such as the lean mass, the water compartment or the fat compartment using bioelectrical impedance analysis
* To define the neurological status by ataxia score
* To get a detailed immune status, vaccination status and liver values as well as special tumor markers in blood
* To check the lung function using spirometry
* To measure liver stiffness using transient elastography (FibroScan)
* To compile any symptoms of infection by diary
* To investigate the ataxia status and physical condition by means of the Five-Times-Sit-to-Stand Test

Visit 2 and 4 are additionally conducted as study visits:

* To get a detailed immune status in blood
* To check the lung function using spirometry

ELIGIBILITY:
Inclusion Criteria:

* aim group: genetically and/or clinically diagnosed A-T
* age 2-45 years
* written informed consent

Exclusion Criteria:

* age < 2 or > 45 years
* other diseases with influence on the immune system (i.e. diabetes mellitus, malignoma, dialysis-dependent renal failure)

Ages: 2 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-10-01 (Actual); Primary Completion 2018-09-30 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Infections in A-T | 24 months
  Evaluation of frequency, severity and intensity of infections in A-T patients with and without immunoglobulin G substitution

SECONDARY OUTCOMES:
Liver disease | 24 months
  Evaluation of the degree of liver disease measured by liver enzymes and structural changes by transient elastography (Fibroscan) in A-T patients
Cancer risk | 24 months
  Evaluation of tumor markers in A-T patients

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Zielen, Prof. Dr., Principal Investigator — Children's Hospital, Allergology, Pneumology and Cystic Fibrosis, Goethe-University
Locations (1):
- Children's Hospital, Allergology, Pneumology and Cystic Fibrosis, Goethe University Frankfurt, Frankfurt am Main, Hesse, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zielen S, Duecker RP, Woelke S, Donath H, Bakhtiar S, Buecker A, Kreyenberg H, Huenecke S, Bader P, Mahlaoui N, Ehl S, El-Helou SM, Pietrucha B, Plebani A, van der Flier M, van Aerde K, Kilic SS, Reda SM, Kostyuchenko L, McDermott E, Galal N, Pignata C, Perez JLS, Laws HJ, Niehues T, Kutukculer N, Seidel MG, Marques L, Ciznar P, Edgar JDM, Soler-Palacin P, von Bernuth H, Krueger R, Meyts I, Baumann U, Kanariou M, Grimbacher B, Hauck F, Graf D, Granado LIG, Prader S, Reisli I, Slatter M, Rodriguez-Gallego C, Arkwright PD, Bethune C, Deripapa E, Sharapova SO, Lehmberg K, Davies EG, Schuetz C, Kindle G, Schubert R. Simple Measurement of IgA Predicts Immunity and Mortality in Ataxia-Telangiectasia. J Clin Immunol. 2021 Nov;41(8):1878-1892. doi: 10.1007/s10875-021-01090-8. Epub 2021 Sep 3. PMID 34477998